CLINICAL TRIAL: NCT06270472
Title: Trans Inguinal Periperitoneal Technique in Inguinal Hernioplasty at General Surgery Department in Assiut University Hospitals
Brief Title: Transinguinal Periperitoneal Technique in Inguinal Hernioplasty
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Mohamed Elsayed, Principal Investigator, Assiut University
Other Study IDs: tipp technique
Record Dates: First submitted 2023-12-20; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hernioplasty — The polysome repair was carried out as described by pelisse . In the case of a lateral hernia, the spermatic cord was mobilised and the cremasteric fibers were separated (in men). The hernia sac was dissected from the cord structures and reduced in the preperitoneal space through the internal ring. A dissection gauze was inserted through the internal ring to create the preperitoneal space. The medial border of the internal ring and the epigastric vessels were lifted with a refractor and blunt digital dissection was carried out in the preperitoneal space in all directions. A pocket was created to allow a complete expansion of the mesh. The conventional mesh was introduced with blunt forceps and, after the gauze has been removed, positioned in the preperitoneal space .
  In the case of a medial hernia, the preperitoneal space was reached by incising the transversalis fascia around the base of the sac. Completion of the repair is the same as the lateral hernia procedure.

SUMMARY:
evaluation of feasibility and efficacy of trans inguinal periperitoneal technique by using conventional mesh inguinal hernia repair in general surgery department in Assiut university hospitals

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most commonly performed surgical procedures worldwide with approximately 20 million cases every year . The open Lichtenstein tension-free hernioplasty is most commonly performed and recognized for its low recurrence rate and short learning curve, but associated with an undesirably high level of postoperative chronic groin pain, up to 10-35% . Therefore, chronic groin pain is a common concern after inguinal hernia surgery. Treatment of chronic groin pain can be challenging and may require several interventions including, local anaesthesia , corticosteroids or additional surgery . Several studies showed that chronic groin pain might be dependent on the surgical technique, including identification and handling of inguinal nerves ,Preperitoneal techniques like the transinguinal preperitoneal patch (TIPP )have been developed to minimize these risks. The TIPP technique which introduced by prissier involves a standard anterior inguinal approach, with high dissection and preperitoneal reduction use of a PolySoft mesh have been proved to cause less chronic pain than the Lichtenstein technique. The PolySoft mesh is a lightweight polypropylene mesh, tailored in asymmetric oval shape that contains a recoil ring. Recent studies deficient in evaluation feasibility and efficacy of trans inguinal periperitoneal technique by using conventional mesh in inguinal hernia repair . So the aim of our study to evaluate the use of conventional mesh in transinguinal preperitoneal technique in inguinal hernioplasty .

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years
* fit for surgery.

Exclusion Criteria:

* Patients less than 18 years
* American Society of Anesthesiologists (ASA) 3 : a patient with severe systemic disease as ( poorly treated hypertension or diabetes , morbid obesity , chronic renal failure , stable angina & implanted pacemaker ) .

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. Patients more than 18 years
  2. fit for surgery. 1-Patients less than 18 years 2- ASA 3 : a patient with severe systemic disease as ( poorly treated hypertension or diabetes , morbid obesity , chronic renal failure , stable angina & implanted pacemaker
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of inguinal hernia 2 years follow up . | 2 years
  Recurrence rate of inguinal hernia 2 years follow up .
Numerical rating score of pain | 1year
  Uses numbers to rate postoperative pain

REFERENCES:
- [Background] Messias BA, Almeida PL, Ichinose TMS, Mocchetti ER, Barbosa CA, Waisberg J, Roll S, Ribeiro Junior MF. The Lichtenstein technique is being used adequately in inguinal hernia repair: national analysis and review of the surgical technique. Rev Col Bras Cir. 2023 Dec 8;50:e20233655. doi: 10.1590/0100-6991e-20233655-en. eCollection 2023. PMID 38088634
- [Background] Damous SHB, Damous LL, Borges VA, Fontella AK, Miranda JDS, Koike MK, Saito OC, Birolini CAV, Utiyama EM. Bilateral inguinal hernia repair and male fertility: a randomized clinical trial comparing Lichtenstein versus laparoscopic transabdominal preperitoneal (TAPP) technique. Surg Endosc. 2023 Dec;37(12):9263-9274. doi: 10.1007/s00464-023-10499-8. Epub 2023 Oct 25. PMID 37880447
- [Background] Shekouhi R, Farz F, Sohooli M, Mohammadi S, Abbasi A, Razaghi M, Fereydouni M, Sohrabi M, Seyed-Alagheband SA, Darabi MH. Investigating the safety and efficacy of nerve stimulation for management of groin pain after surgical herniorrhaphy: a systematic review and meta-analysis. Hernia. 2023 Dec;27(6):1363-1373. doi: 10.1007/s10029-023-02861-5. Epub 2023 Aug 19. PMID 37597107